CLINICAL TRIAL: NCT05432037
Title: Evaluation of Cultural Adaptation and Psychometric Properties of Urdu Version of Fear Avoidance Belief Questionnaire
Brief Title: Urdu Version of Fear Avoidance Belief Questionnaire: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00245
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: Fear Avoidance Belief Questionnaire; Urdu Version; Reliability; Validity; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to translate and culturally adapt Fear Avoidance Belief Questionnaire into the Urdu language and to investigate the reliability and validity in the Pakistani population and check its correlation with Visual Analog Scale , Ronald Morris Questionnaire, Quebec Back Pain Disability Scale and Hospital Anxiety and Depression scale .

DETAILED DESCRIPTION:
As per preceding commendation, Fear Avoidance Belief Questionnaire will be translated into Urdu language from its English version and adapted culturally in Pakistan. Among low back pain population, Fear Avoidance Belief Questionnaire will be conducted in 180 patients recruited by convenience sampling technique under the pre-defined inclusion and exclusion criteria after signing consents forms. For testing inter-observer reliability and intra-observer reliability of Fear Avoidance Belief Questionnaire, Hospital anxiety and depression scale, Ronald Morris questionnaire, Quebec pain rating scale and numeric pain rating scale will be administrated by two observers, on the same day, with a time interval of 2 hours between 1st and 2nd conduction. As for the 3rd conduction, it will be carried out after seven days by the first observer, for intra-observer assessment. Statistical Package of Social Sciences software version 24 will be used for the purpose of data entry and analysis. Internal consistency will be assessed by using an intra-class correlation coefficient. The Fear Avoidance Belief Questionnaire will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients or the ones next to them who gave informed consent
* Participants with complain of low back pain for more than 3 months.
* Age at least above 18 years.

Exclusion Criteria:

* Inability to understand or follow the instructions of the Fear Avoidance Belief Questionnaire.
* Any musculoskeletal pathologies
* Suffering from any cardiovascular pathologies
* Any history of tumor and cancer
* Any history of fracture
* Any histories of infections
* Any history of neurological disorders
* Having any spinal deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population for this study will be reported cases of low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Fear Avoidance Belief Questionnaire | 1st day
  The fear avoidance belief questionnaire is a standardized clinical assessment tool to investigate patients work and activity specific fear-avoidance beliefs and physical disability related to work. The Fear Avoidance Belief Questionnaire consists of 2 sub-scales. The Physical Activity sub-scale and The Work sub-scale.
Hospital Anxiety and Depression scale | 1st day
  It is the scale used for evaluation of anxiety and depression symptoms related to disease. The Hospital Anxiety and Depression scale is the objective assessment of disease related anxiety and depression symptoms based on 14 items. 7 questions for each depression and anxiety sub-scales.
  Scoring ranges from 0-3. Total scores are from 0-21. Normal or no anxiety scores from 0-7, 8-10 mild to moderate anxiety, 11-21 moderate to severe anxiety.
Ronald Morris Questionnaire | 1st day
  Ronald Morris Questionnaire is the scale used for evaluation of level of disability among patients of back pain. Ronald Morris questionnaire is a self-administrated disability measurement based on 24 items. Higher level of disability is represented by greater score on 24-points scale.
Quebec Pain Rating Scale | 1st day
  The Quebec Back Pain Disability Scale is a 20-item self-administered device designed to assess the level of practical disability in people with low back pain. The scale is a reliable and accurate measure used to monitor the progress of individual patients participating in treatment or rehabilitation programs.
Visual Analog Scale | 1st day
  Scores of Visual Analog Scale are based on self-reported measures of symbols that are recorded with a length of 10 as well as a written mark placed in one place. The centimetre line that represents the continuity between the two ends of the scale - from "no pain" on the left end of the scale (0 cm) and the "worst pain" on the right end of the scale (10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No